CLINICAL TRIAL: NCT04953702
Title: Insufficiency Fractures of the Knee: Insufficient of Nutrients or Cartilage?
Brief Title: Study of the Associations Between Subchondral Insufficiency Fractures of the Knee and Pre-existing Health, Lifestyle, and/or Musculoskeletal Conditions
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial/IRB Approval Lapsed
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: H00023240
Record Dates: First submitted 2021-06-11; First posted 2021-07-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Subchondral Insufficiency Fracture
Keywords: Exercise; Musculoskeletal diseases; Nutrition disorders; Pain
MeSH Terms: conditions — Motor Activity; Musculoskeletal Diseases; Nutrition Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study is designed to investigate possible association(s) between subchondral insufficiency fractures (SIFKs) of the knee and pre-existing health, lifestyle, and/or musculoskeletal conditions. In doing so, this research may shed light on the underlying cause(s) of SIFKs. It is hypothesized that SIFKs of the knee are related to osteoarthritis, weak bone, and/or metabolic issues, rather than trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SIFK from ages ≥18 years old who seek treatment at the University of Massachusetts for their musculoskeletal care.

Exclusion Criteria:

* Patients with a history of associated conditions such as cancer, inflammatory arthritis, or chronic alcohol or tobacco dependence will be excluded.

The following special populations will be excluded:

* Adults unable to consent and/or unable to follow two-step commands
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Non-English-speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with SIFK from ages ≥18 years old who seek treatment at the University of Massachusetts for their musculoskeletal care and are not a member of a special population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Correlation between subchondral insufficiency fractures (SIFKs) and coexisting conditions | 12 months
  The proportion of patients with subchondral insufficiency fractures and coexisting conditions (overall and per condition) as compared to those without coexisting conditions.
  Coexisting conditions are identified and defined through metabolic and musculoskeletal-related findings from available lab and radiological results in the patient medical record, such as those related to diabetes, obesity, osteoarthritis and other orthopedic related conditions and metabolic issues.

SECONDARY OUTCOMES:
Correlation between type of treatment for subchondral insufficiency fractures (SIFKs) and treatment outcome (pain level) | 12 months
  The proportions of patients with improvement in pain, worsening of pain, or no change in pain per prescribed treatment.
  Changes in pain level identified by visual analog scale (VAS) and three-point scale (same/better/worse). The VAS includes subject identification of pain level from 0 (no pain) to 10 (worst pain). Change in pain level identified via VAS in evaluating numerical assessment provided by subjects over course of treatment (increase in rank = worsening; decrease in rank = improving; same rank = same). Change in pain level identified directly using the three point scale (same/better/worse).
Correlation between activity level and treatment outcome (pain level) | 12 months
  The proportions of patients with improvement in pain, worsening of pain, or no change in pain based on activity level.
  Changes in pain level identified by visual analog scale (VAS) and three-point scale (same/better/worse). The VAS includes subject identification of pain level from 0 (no pain) to 10 (worst pain). Change in pain level identified via VAS in evaluating numerical assessment provided by subjects over course of treatment (increase in rank = worsening; decrease in rank = improving; same rank = same). Change in pain level identified directly using the three point scale (same/better/worse).
  Activity level collected via interviews (exercise type/duration/frequency). Activity level categorized into none/mild/moderate/high exertion based on the following criteria:
  * MILD=pool, chair yoga, golf w/ cart
  * MODERATE=land-based exercise/standing/walking/cycling, golf w/out cart
  * HIGH=can't talk while exercising, running/cycling>10miles, jumping, boot camp
Correlation between coexisting conditions and treatment outcome (pain level) | 12 months
  The proportions of patients with improvement in pain, worsening of pain, or no change in pain based on presence or absence of coexisting conditions (overall, per condition).
  Changes in pain level identified by visual analog scale (VAS) and three-point scale (same/better/worse). The VAS includes subject identification of pain level from 0 (no pain) to 10 (worst pain). Change in pain level identified via VAS in evaluating numerical assessment provided by subjects over course of treatment (increase in rank = worsening; decrease in rank = improving; same rank = same). Change in pain level identified directly using the three point scale (same/better/worse).
  Coexisting conditions identified and defined through metabolic and MSK-related findings from available lab and radiological results in the medical record, such as those related to diabetes, obesity, osteoarthritis and other orthopedic related and metabolic issues.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Scarpetti, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Memorial Health, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No